CLINICAL TRIAL: NCT04116099
Title: An Observational Registry Evaluating the Flexitouch® Plus in Vascular Clinic Patients With Lower Extremity Lymphedema
Brief Title: CVR Registry Evaluating Flexitouch Plus and Conservative Care vs Conservative Care Only for Treatment of Lymphedema
Status: Terminated | Type: Observational
Why Stopped: Covid impact - slow enrollment
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 5020
Record Dates: First submitted 2019-09-11; First posted 2019-10-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Lymphedema
Keywords: Lymphedema of Leg; Chronic Venous Insufficiency; Primary Lymphedema; Secondary Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Conservative care alone: Conservative care alone which may include graduated compression, manual lymphatic drainage (MLD) performed by a licensed therapist, self-MLD, and instruction on exercise and skin care.
  Interventions: Other: Conservative care
- Flexitouch Plus and conservative care: Flexitouch Plus and conservative care which includes Flexitouch Plus treatment as well as conservative care measures which may include graduated compression, manual lymphatic drainage (MLD) performed by a licensed therapist, self-MLD, and instruction on exercise and skin care.
  Interventions: Other: Conservative care; Device: Flexitouch Plus

INTERVENTIONS:
Other: Conservative care — May include graduated compression, MLD performed by a licensed therapist, self-MLD, and instruction on exercise and skin care.
Device: Flexitouch Plus — Flexitouch Plus treatment.
  Groups: Flexitouch Plus and conservative care

SUMMARY:
Subjects with lower extremity lymphedema will be prescribed, per standard of care, to either Flexitouch Plus with conservative care or conservative care only and be followed for 12 months.

DETAILED DESCRIPTION:
Conservative care treatment for lymphedema may include use of compression, manual lymphatic drainage (MLD, performed either by a therapist or self-MLD), exercises and skin care. Subjects presenting to a vein clinic (Center for Vein Restoration or CVR) with lymphedema of the lower extremity/ies may receive a standard-of-care prescription for conservative care or for the Flexitouch Plus pneumatic compression device along with conservative care. Subjects will be followed (by phone and in clinic) for 12 months after initiating treatment for venous- and lymphedema-related complications, unscheduled visits, changes in quality of life measures and edema measures, skin changes, and changes to wounds (if present).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older.
2. Diagnosis of lower extremity lymphedema (including primary, secondary, chronic venous insufficiency (CVI)-related, unilateral, or bilateral).
3. Clinical Etiology Anatomy Pathophysiology (CEAP) Classification of C3 or higher.
4. Willing to comply with prescribed care, protocol requirements, and study-related visits.
5. Willing and able to provide consent to participate.

Exclusion Criteria:

1. BMI > 50.
2. Significant venous reflux disease, as determined by the investigator (e.g., indicated for venous intervention, post intervention with inadequate venous function, or ultrasound evidence of deep venous obstruction).
3. Unresolved healing at the surgical site following a venous intervention (e.g., ablation, stenting, or venoplasty).
4. Heart failure (acute pulmonary edema, decompensated acute heart failure).
5. Acute venous disease (< 6 weeks) such as acute thrombophlebitis, acute deep venous thrombosis, or acute pulmonary embolism.
6. Significant peripheral artery disease (ankle-brachial index (ABI) < 0.6, critical limb ischemia including ischemic rest pain, arterial wounds or gangrene).
7. Active skin or limb infection/ inflammatory disease (acute cellulitis, other uncontrolled skin or untreated inflammatory skin disease).
8. Active cancer (cancer that is currently under treatment, but not yet in remission).
9. Poorly controlled kidney disease (glomerular filtration rate < 30 mls per minute), hypoproteinemia, pulmonary hypertension, hypothyroidism, cyclic edema, or Munchausen Syndrome.
10. Any circumstance where increased lymphatic or venous return is undesirable.
11. Currently pregnant or trying to become pregnant (for Flexitouch Plus and conservative care group).
12. Current participation in any drug or other device clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be drawn from vascular patients with lower extremity lymphedema that is unilateral or bilateral.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Complications | 12 months
  To evaluate the Flexitouch Plus and conservative care, compared to conservative care alone, in vascular patients with lower extremity lymphedema after 12 months of treatment based upon the number of lymphedema and venous-related complications.
Number of unscheduled visits | 12 months
  To evaluate the Flexitouch Plus and conservative care, compared to conservative care alone, in vascular patients with lower extremity lymphedema after 12 months of treatment based upon the number of lymphedema and venous-related unscheduled follow-up visits (non-routine clinic, hospital, urgent care, and emergency room visits).

SECONDARY OUTCOMES:
Quality of life changes: Short-Form 12 (SF-12) | 6 months
  To evaluate the effectiveness of the Flexitouch Plus and conservative care, compared to conservative care alone, in vascular patients with lower extremity lymphedema after 6 months of treatment based upon changes in the SF-12. This survey includes 12 questions to measure physical and mental health from the patient's point of view. The questionnaire includes eight health domains: physical functioning, physical health problems, bodily pain, general health, vitality, social functioning, emotional health problems, and mental health. The scoring mechanism uses T scores for all surveys using means and standard deviations from the 1998 US general population. A higher score represents better function.
Quality of life changes: Quality of Life with Venous Insufficiency (CIVIQ-20) | 6 months
  To evaluate the effectiveness of the Flexitouch Plus and conservative care, compared to conservative care alone, in vascular patients with lower extremity lymphedema after 6 months of treatment based upon changes in the CIVIQ-20, which is a survey specific to assess patient-perceived quality of life with chronic venous disorders. The instrument reviews four dimensions - psychological (range 9-45), pain (range 4-20), physical (range 4-20), and social (range 3-15). A global index score can be obtained by adding up the scores of all 20 items (range 20-100). A low score corresponds to greater patient comfort.
Quality of life changes: Lymphedema Quality of Life Tool (LYMQOL) | 6 months
  To evaluate the effectiveness of the Flexitouch Plus and conservative care, compared to conservative care alone, in vascular patients with lower extremity lymphedema after 6 months of treatment based upon changes in the LYMQOL, used to assess lymphedema symptom changes. LYMQOL includes sub-scores for function (range 8-32), appearance (range 7-28), symptoms (range 5-20), and mood (range 6-24) where lower scores represent a better outcome. It also includes an overall QOL sub-score (range 0-10) where a higher score represents a better outcome.
Quality of life changes: Clinical Global Impression of Change - Global Improvement (CGI-I) | 6 months
  To evaluate the effectiveness of the Flexitouch Plus and conservative care, compared to conservative care alone, in vascular patients with lower extremity lymphedema after 6 months of treatment based upon a clinician's response to one question at the 6 month follow-up visit pertaining to overall clinical improvement (range 1-7). A lower score signifies greater improvement.
Quality of life changes: Patient Global Impression of Change (PGIC) | 6 months
  To evaluate the effectiveness of the Flexitouch Plus and conservative care, compared to conservative care alone, in vascular patients with lower extremity lymphedema after 6 months of treatment based upon the patient's response to one question at the 6 month follow-up visit pertaining to overall status change (range 1-7). A lower score signifies greater improvement.
Edema measures | 6 months
  To evaluate the effectiveness of the Flexitouch Plus and conservative care, compared to conservative care alone, in vascular patients with lower extremity lymphedema after 6 months of treatment based upon changes in edema measures on affected/ most affected leg.
Presence and severity of skin changes | 6 months
  To evaluate the effectiveness of the Flexitouch Plus and conservative care, compared to conservative care alone, in vascular patients with lower extremity lymphedema after 6 months of treatment based upon skin changes on affected/ most affected leg.
Wound area | 6 months
  To evaluate the effectiveness of the Flexitouch Plus and conservative care, compared to conservative care alone, in vascular patients with lower extremity lymphedema after 6 months of treatment based upon percent wound area reduction in subjects presenting with wounds.

OTHER OUTCOMES:
Flexitouch Plus treatment satisfaction | 6 months
  To evaluate Flexitouch Plus treatment satisfaction after 6 months of treatment.
Call volume | 12 months
  Assess subject call volume for conservative care subjects compared to subjects using the Flexitouch Plus and conservative care.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pappas, Principal Investigator — Center for Vein Restoration
Locations (3):
- United States (3):
  - Center for Vein Restoration - Glen Burnie, Glen Burnie, Maryland
  - Center for Vein Restoration - Greenbelt, Greenbelt, Maryland
  - Center for Vein Restoration - Silver Spring, Silver Spring, Maryland

IPD SHARING:
Plan to Share IPD: No